CLINICAL TRIAL: NCT00336778
Title: A Phase I Pilot Study Of An Antiretroviral Bridging Regimen In Highly Experienced Patients Unable To Achieve Viral Suppression.
Brief Title: Phase 1 Pilot Study of an ART Bridging Regimen in Highly Experienced Patients Unable to Achieve Viral Suppression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22675
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 3TC, TDF, NLV — 3TC 300 mg PO once daily+ TDF 300 mg PO once daily+ NLV 1250 mg PO twice daily (after 12 week lead-in period)

SUMMARY:
We hypothesize that a simple bridging ARV regimen that tends to select for virus with a low replicative capacity may tend to stabilize CD4 cell counts and HIV viral load and might be an option to consider in patients with MDR HIV.

This strategy will provide them with the bridge they desperately need so that they can await the development of new therapies that when used in combination will give them the best chance in achieving complete virologic suppression.

DETAILED DESCRIPTION:
Bridge is a pilot, single-arm, open-label, study to assess the ability of 3 FDA approved anti-retroviral drugs to decrease replication capacity of HIV virus in order to stabilize CD4 cell count and HIV RNA viral loads . All subjects will be prescribed the three-drug combination of lamivudine (3TC) + tenofovir disoproxil fumarate (TDF) + nelfinavir (NLV)The "Bridge Study" is a pilot, study to assess the ability of 3 FDA approved anti-retroviral drugs to decrease replication capacity of HIV virus in order to stabilize CD4 cell count and HIV RNA viral loads. All subjects will receive the three-drug combination of lamivudine (3TC)+tenofovir disoproxil fumarate(TDF)+nelfinavir (NLV)

The study will enroll 12 subjects for a 48 week study. Major entry criteria include: HIV+ Men and women 18 years of age who are currently failing antiretroviral(ARV)therapy with an HIV-1 RNA VL > 10,000 and have failed multiple treatment regimens due to resistance and/or intolerance. Genotype must demonstrate resistance to 3 major classes of ARV's - PI's, NNRTI's, and NRTI's.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age > 18 years of age.
2. Ability and willingness to give written informed consent.
3. HIV-1 infection as documented by any licensed ELISA test kit and confirmed by either Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA prior to study entry.
4. Patient failed multiple treatment regimens due to development of viral resistance/and or intolerance.
5. Patient's provider feels that patient has exhausted currently available treatment options and that it is highly unlikely that a regimen (including one that contains T-20) could be constructed that would result in sustained virologic suppression at this time.
6. Evidence of MDR virus (broad 3 class resistance) based on the results of the MDR-HIV qualifying screening genotypic resistance test or a history of a previous genotypic resistance test.
7. The following screening laboratory values obtained within 30 days prior to study entry:

   * HIV-1 RNA or BDNA > 10,000 copies/mL

Exclusion Criteria:

1. Active drug or alcohol abuse or dependence which, in the opinion of the investigator, would interfere with adherence to study requirements.
2. History of any illness that, in the opinion of the study investigators, might confound the results of the study or pose additional risk in administering study drugs to the subject.
3. Acute therapy for a serious infection or other serious medical illnesses that are potentially life threatening and require systemic therapy and/or hospitalization.

   NOTE: Subjects with a serious infection or serious medical illness must complete acute therapy at least 7 days prior to study entry. Subjects with all other infections or medical illnesses (e.g., vaginitis, folliculitis, bronchitis, pharyngitis, thrush) must receive appropriate therapy prior to study entry (no time restriction).
4. Significant Renal Insufficiency - calculated creatinine clearance < 50
5. Upon reviewing medication history and genotypic resistance testing, study investigators feel that would be inappropriate to enroll patient in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in replication capacity over time from baseline to week 48. | 48 weeks
  Change in viral replication capacity

SECONDARY OUTCOMES:
Change in viral load from baseline to week 48. | 48 weeks
  Change in viral load
Change in CD4 cell count from baseline to week 48. | 48 weeks
  Change in CD4
Time to first Grade 3 sign, symptom, or lab abnormality,and/or OI that is at least a grade higher than baseline or a significant increase in viral load from baseline or a greater than 50% decline in CD4 cell count | 48 weeks
  Grade 3 sign, symptom, lab abnormality, OI that has exacerbated. Or a significant increase in viral load from baseline or a greater than 50% decline in CD4

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Redfield, MD, Study Director — University of Maryland, College Park
Locations (2):
- United States (2):
  - University of Maryland Baltimore, Institute of Human Virology, Baltimore, Maryland
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland